CLINICAL TRIAL: NCT05359965
Title: Effect of Continuous Positive Airway Pressure (CPAP) on Abnormal Gastroesophageal Reflux and Lung Inflammation in Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Effect of CPAP on Abnormal Gastroesophageal Reflux and Lung Inflammation in IPF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IIS2018-10747
Record Dates: First submitted 2022-02-21; First posted 2022-05-04 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Pulmonary Fibrosis; Obstructive Sleep Apnea; Gastro Esophageal Reflux
Keywords: IPF; OSA; GERD
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Sleep Apnea, Obstructive; Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to treatment groups using a 1:1 randomized block design via the randomization module in REDCap. The PI and study coordinator will be blinded to next assignment.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Study investigators and care providers will be blinded and not involved in any CPAP or no CPAP related set-up, instruction, or device troubleshooting during the course the treatment phase. Lab personnel performing biomarker analysis will only have access to subject study ID and not treatment group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CPAP (Experimental): Subjects randomized to the treatment arm, will receive continuous positive airway pressure (CPAP) while sleeping via an autoPAP device for 4-8 weeks.
  Interventions: Device: Positive Airway Pressure
- No CPAP (No Intervention): Subjects assigned to the no CPAP group will not have any intervention for a 4-8 week period.

INTERVENTIONS:
Device: Positive Airway Pressure — Gentle and steady pressure (with or without supplemental oxygen) delivered to the airways of the lungs while subjects are sleeping.
  Arms: CPAP

SUMMARY:
This study will evaluate the effect of CPAP therapy on esophageal pH and lung inflammation in patients with idiopathic pulmonary fibrosis (IPF) and sleep apnea.

DETAILED DESCRIPTION:
Participants in this study will have an overnight sleep study done while wearing a 24 hour pH monitor in the esophagus. If the participant has sleep apnea, he or she will be randomly assigned to receive either CPAP treatment or no CPAP treatment. After 4-8 weeks, the participant will have another overnight sleep study with 24 hour pH monitoring. Blood will also be collected at both time points and again after 6 months to measure biomarkers that are related to lung inflammation.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of IPF based on the 2018 IPF guidelines
* high likelihood of OSA based on the STOP-BANG measure, with a score of 3 or greater
* patients on nintedanib, or in whom nintedanib will be initiated prior to enrollment in the study
* able to participated in 24hr pH monitoring
* able to comply with CPAP treatment
* able to provide written informed consent prior to any study procedures
* willing to complete all study measurements and assessments in compliance with the protocol

Exclusion Criteria:

* interstitial lung disease caused by conditions other than IPF
* severe concomitant illness limiting life expectancy (< 1 year)
* residual lung volume > or equal to 120% of predicted
* obstructive lung disease: FEV1/FVC ratio < 0.70
* current drug or alcohol dependence
* patients who are unable to tolerate nintedanib
* patients who are unable to use CPAP or are unwilling to participate in the 24 hr pH probe placement
* patients who were diagnosed with recent IPF exacerbation within 4 weeks of enrollment (may be rescheduled for enrollment once recovered)
* patients who have had prior nasal surgery or trauma that would make pH probe placement difficult
* patients on anticoagulation (aspirin is not an exclusion)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Composite Biomarker Score | 4-8 weeks
  The primary outcome will be a composite value that is a weighted average of z-scores of the biomarkers MMP1, MMP7, IL-8, KL-6, and CXCL13, weighted by the univariate effect sizes of each biomarker. MMP1, MMP7, IL-8, KL-6, and CXCL13 will be measured using enzyme linked immunosorbent assays (ELISA) for these analytes. (Z-score is a unitless number, as is the weighted average.)

SECONDARY OUTCOMES:
Biomarker of Lung Inflammation: KL-6 | 4-8 weeks
  The value of KL-6 measured by ELISA in U/ml.
Biomarker of Lung Inflammation: MMP1 | 4-8 weeks
  The value of MMP1 measured by ELISA in ng/ml.
Biomarker of Lung Inflammation: MMP7 | 4-8 weeks
  The value of MMP7 measured by ELISA in ng/ml.
Biomarker of Lung Inflammation: IL-8 | 4-8 weeks
  The value of IL-8 measured by ELISA in pg/ml.
Biomarker of Lung Inflammation: CXCL13 | 4-8 weeks
  The value of CXCL-13 measured by ELISA in pg/ml.
Esophageal pH During Sleep | 4-8 weeks
  Total sleep time (in minutes) with pH less than 4.
24hr-Esophageal pH | 4-8 weeks
  Total time (minutes in 24hr period) with pH less than 4.
FVC change | 6 months
  FVC change in percentage of predicted values over 6 months (baseline to 6 months).
Composite Biomarker Score at Six Months | 6 months
  Weighted average of z-scores of the biomarkers MMP1, MMP7, IL8, KL-6, and CXCL13, weighted by the univariate effect sizes of each biomarker at six months. (Z-score is a unitless number, as is the weighted average.)

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Chaudhary, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No